CLINICAL TRIAL: NCT05773326
Title: A Phase 0, Single-center, Open-label, Dose-escalating Trial Using Super-selective Intra-arterial Infusion of a Single Dose of Temsirolimus for the Treatment of Recurrent High-grade Glioma
Brief Title: Superselective Intra-arterial Cerebral Infusion of Temsirolimus in HGG
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Barrow Neurological Institute (Other); Ivy Brain Tumor Center (Other)
Responsible Party: Sponsor-Investigator, Nader Sanai, Director of the Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-17
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: High Grade Glioma; Glioma; Glioma, Malignant; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single infusion of Temsirolimus (Experimental): Single infusion of Temsirolimus via super-selective intra-arterial infusion or IV
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — TORISEL® (temsirolimus) is a kinase inhibitor indicated for the treatment of advanced renal cell carcinoma.
  Other Names: Torisel

SUMMARY:
This is a single-center, open-label, dose-escalating Phase 0 trial that will enroll participants with a confirmed diagnosed recurrent high-grade glioma (grade 3 or 4 per WHO criteria) targeting the mTOR pathway. Eligible participants will be administered a single infusion of temsirolimus through super-selective intra-arterial infusion or intravenous infusion. Participants will receive the study drug administration on the same day as the planned surgical resection of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed high-grade glioma (Grade 3 or 4 per 2021 WHO criteria) in the frontal lobe.
* Tissue must demonstrate mTOR+: PTEN loss OR PIK3C2B or AKT3 amplification on aCGH OR mutations for PIK3CA or PIK3R1, or mTOR or PTEN mutations using next-generation sequencing analysis OR pS6 positivity on immunohistochemistry (≥30% for pS6).
* Patients who have completed the Stupp regimen.
* Have measurable disease pre-operatively, defined as at least 1 contrast enhancing lesion, with 2 perpendicular measurements of at least 1 cm, as per RANO criteria.
* Sufficient biopsy or archival tissue to confirm eligibility
* Has voluntarily agreed to participate by giving written informed consent. Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
* Age ≥18 at time of consent.
* Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology (Group (ECOG) scale
* Participant has adequate bone marrow and organ function
* Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
* For females of reproductive potential: use of highly effective contraception and agreement to use such a method during study participation until the end of treatment administration and for 3 months after the last dose of study drug.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner until the end of treatment administration and for 3 months after the last dose of study drug.
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Pregnancy or lactation.
* Known hypersensitivity to temsirolimus or its metabolites, polysorbate 80, or to any other component of temsirolimus.
* Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, active infection, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance]
* Received a live vaccination or is in close contact with someone who received a live vaccination within 28 days of the start of study treatment
* Treatment with another investigational drug or other intervention within 30 days prior to the planned treatment Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Tumor pharmacokinetics (PK) of temsirolimus | Day 1 (Intraoperative)
  Total and unbound temsirolimus concentration in tumor tissue.

SECONDARY OUTCOMES:
Pharmacodynamic effects of temsirolimus | Day 1 (Intraoperative)
  Quantification of the % of pS6 positive cells

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Chief Scientific Officer/Director
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ivy Brain Tumor Center Website — http://ivybraintumorcenter.org